CLINICAL TRIAL: NCT03602820
Title: A Long-Term Follow-Up Study in Subjects Who Received an Adenovirus-Associated Viral Vector Serotype 2 Containing the Human RPE65 Gene (AAV2-hRPE65v2, Voretigene Neparvovec-rzyl) Administered Via Subretinal Injection
Brief Title: Long-term Follow-up Study in Subjects Who Received Voretigene Neparvovec-rzyl (AAV2-hRPE65v2)
Status: Active, not recruiting | Type: Observational
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AAV2-hRPE65v2-LTFU-01
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Inherited Retinal Dystrophy Due to RPE65 Mutations
Keywords: Leber congenital amaurosis, retinitis pigmentosa
MeSH Terms: conditions — Leber Congenital Amaurosis; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: AAV2-hRPE65v2
  Other Names: Voretigene Neparvovec-rzyl

SUMMARY:
Multi-site, non-randomized, observational study, for up to 15 years after subretinal AAV2-hRPE65v2 administration for each subject. The study is a non-interventional, follow-up study of subjects who participated in previous AAV2-hRPE65v2 gene therapy clinical trials.

DETAILED DESCRIPTION:
This is an observational follow-up study of subjects who participated in previous Phase 1 and Phase 3 clinical trials of AAV2-hRPE65v2 gene therapy (voretigene neparvovec-rzyl) to evaluate long term durability and safety for 15 years after subretinal administration.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who participated in prior subretinal AAV2-hRPE65v2 gene therapy clinical studies

Exclusion Criteria:

1. Subjects who will not consent for study.
2. Subjects who the investigators believe are not capable of performing study assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who received the subretinal administration of AAV2-hRPE65v2 (voretigene neparvovec-rzyl) in the Phase 1 or Phase 3 clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Mobility testing, Bilateral | 15 years
  Mobility testing will be videotaped at each study visit at which it is conducted. Independent reviewers may grade subjects' mobility videos. Graders will use a defined combination of speed and accuracy to grade each course attempt at a given light intensity. The course will be re-configured between each attempt, using twelve standardized templates, to reduce the impact of a potential learning effect. Each subject will be tested, using both eyes, under at least two and sometimes three different (specified) lighting conditions. The levels of light, selected to span lighting conditions that individuals encounter in daily life, range from a studio with floodlights (400 lux) or a brightly lit office (250 lux) down to a poorly lit sidewalk at night (1 lux).

SECONDARY OUTCOMES:
Full-field light sensitivity threshold (FST) testing | 15 years
  FST testing measures the light sensitivity of the entire visual field by recording the luminance at which a subject reports seeing the dimmest flash. The test is carried out on subjects with dilated eyes in a dark-adapted state; subjects are seated in front of a Ganzfeld dome in which the light flashes are generated. The light sensitivity of each eye is measured separately by patching one eye (and then the other). A sound is generated and the subject presses one button when they see a flash or a second button if they do not see a flash. Flashes of varying luminance (in a range spanning ~80 dB) are presented in a randomized order with no flashes, except that the series starts with dim flashes. From this data, an algorithm calculates the minimum luminance (for each eye) at which the subject perceives light.
Mobility testing, Monocular | 15 years
  Mobility testing will be videotaped at each study visit at which it is conducted. Independent reviewers may grade subjects' mobility videos. Graders will use a defined combination of speed and accuracy to grade each course attempt at a given light intensity. The course will be re-configured between each attempt, using twelve standardized templates, to reduce the impact of a potential learning effect. Each subject will be tested, using the first treated eye, under at least two and sometimes three different (specified) lighting conditions. The levels of light, selected to span lighting conditions that individuals encounter in daily life, range from a studio with floodlights (400 lux) or a brightly lit office (250 lux) down to a poorly lit sidewalk at night (1 lux).
Visual acuity | 15 years
  Visual acuity measures central vision using the ability to resolve standard optotype images presented as letters corresponding to different visual angles, i.e., image size. This testing will include age-adapted tests, such as ETDRS testing or HOTV testing (which uses the letters H, O, T, V, which can be identified even by young children and all four of which center around a vertical axis). The level of central visual resolution is converted to a visual angle score (LogMAR). Subjects may, in some cases, need to undergo repeated testing sessions, including on successive days, to establish consistent measurements on psychophysical tests, such as visual acuity.

OTHER OUTCOMES:
Visual field testing - Humphrey and/or Goldmann | 15 years
  Visual field parameters will evaluate alterations in function of different regions of the retina; kinetic fields will be measured with Goldmann perimetry and static fields with Humphrey computerized testing.
Visual function questionnaire | 15 years
  The gene therapy study investigators developed a questionnaire relevant to the deficit experienced by patients with RPE65 gene mutations. This patient-reported outcome consists of 25 questions pertaining to activities of daily living that are dependent upon vision or have a vision component. Subjects and/or their parent or guardian will be asked to provide all responses regarding the perceived degree of difficulty of these activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Maguire, MD, Principal Investigator — University of Pennsylvania; Stephen Russell, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No